CLINICAL TRIAL: NCT06744075
Title: Study of the Clearance of Minimal Residual Disease Measured at the End of First-line Treatment in Patients Treated for B-cell Lymphoma or Hodgkin Lymphoma
Brief Title: Study of the Clearance of Minimal Residual Disease Measured at the End of First-line Treatment in Patients With Lymphoma
Acronym: CELERITY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHB24.02
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: B-cell Lymphoma; Hodgkin Lymphoma
Keywords: Lymphoma; Liquid biopsy; Minimal Residual Disease; Poitron Emission Tomography; Circulating Tumor DNA
MeSH Terms: conditions — Lymphoma, B-Cell; Hodgkin Disease; Lymphoma; Neoplasm, Residual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CELERITY Arm (Other): CT DNA Collection at baseline, mid-treatment and at the end of treatment
  Interventions: Other: Blood assessment

INTERVENTIONS:
Other: Blood assessment — ctDNA collection (venous blood draw) will occur at baseline, mid-treatment, and at the end of treatment

SUMMARY:
This study aims to assess the feasibility of predicting patient outcomes at 1 year and 2 years after the end of first-line treatment using "liquid biopsy" (monitoring of circulating tumor DNA, ctDNA), compared to the currently recommended examination, which is Positon Emission Tomography (PET-CT) imaging at the end of first-line treatment (assessment of therapeutic response using the Deauville score according to the Lugano 2014 criteria). The study will focus on demonstrating the ability of ctDNA clearance to predict 1-year and 2-year outcomes (lymphoma progression or death) in patients treated with first-line therapy for B-cell lymphoma or Hodgkin lymphoma. This could contribute to establishing minimal residual disease clearance as a key endpoint for evaluating the efficacy of therapeutic strategies in future clinical trials and guiding patient management (e.g., de-escalation or intensification strategies, redirection toward immunotherapy, and theranostic approaches).

DETAILED DESCRIPTION:
Over the past decade, molecular biology methods known as "liquid biopsy" tools have emerged to identify tumor genotypes without a traditional biopsy, using blood samples and sequencing of circulating tumor DNA (ctDNA). Evidence supporting ctDNA's ability to perform comprehensive tumor genotyping, serving as an accurate reflection of the tumor genotype, has been well-documented in the literature. Two key aspects of the clinical relevance and routine applicability of ctDNA are currently under investigation:

The potential to measure and monitor the clearance of minimal residual disease (MRD) during and after treatment, which heavily depends on the detection limit and sensitivity of the analytical method.

The ability to deliver ctDNA analysis results to clinicians in real time, within timelines compatible with patient decision-making.

At Rouen, the investigators now use a method based on Unique Molecular Identifiers (UMIs), a type of molecular barcode that provides increased precision during sequencing. These molecular barcodes are short sequences used to uniquely label each DNA molecule in a sample library, minimizing false positives caused by random sequencing errors. By incorporating individual barcodes into each original DNA fragment, true variants in the original sample can be distinguished from errors introduced during library preparation, target enrichment, or sequencing.

The investigators have developed a new Next Generation sequencing (NGS) panel dedicated to ctDNA analysis using UMIs, encompassing 101 genes and 133 Kb of sequencing regions with phased variants on an Illumina® pipeline.

The panel offers several advantages:

It includes exons of genes involved in lymphomagenesis, with prognostic significance, or that aid in lymphoma classification.

It targets non-coding regions affected by AID (somatic hypermutation). It covers regions frequently impacted by deletions or amplifications (gene copy number variations).

It employs a genomic region capture technique, which, unlike amplicon-based methods, enables the study of the fragmentome. This is important as ctDNA fragmentation profiles are not uniform and may reflect transcriptional and epigenetic changes in the lymphoma's cell of origin, providing additional insights beyond the mutation and somatic variant data commonly used in molecular biology techniques.

The investigators aim to use this panel to refine patient outcome predictions in lymphomas at the end of first-line treatment, with a particular focus on ctDNA kinetics and clearance compared to PET-CT imaging and the synergy between these tools. The investigators anticipate that these findings will support the personalization of therapeutic strategies for lymphoma patients through appropriate escalation or de-escalation approaches guided by MRD. The results of this study will provide the proof of concept necessary for adopting this MRD monitoring test into routine clinical practice for lymphoma patients.

This MRD clearance tracking test could also serve as a key tool in clinical trials for new drug development. By eliminating the need for long follow-up periods required to establish progression-free survival (PFS), this approach could enable earlier interim analyses of efficacy, potentially accelerating and shortening the duration of Phase 3 trials and the clinical development of new lymphoma treatments. If accepted by the academic community as an early efficacy endpoint and a surrogate marker for PFS, this test could significantly impact the design of future lymphoma trials.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Diagnosed with large B-cell lymphoma (including T-cell/histiocyte-rich B-cell lymphoma, high-grade B-cell lymphoma, primary mediastinal B-cell lymphoma), follicular B-cell lymphoma (all grades), mantle cell lymphoma (all variants), marginal zone B-cell lymphoma, or Hodgkin lymphoma (classical Hodgkin lymphoma or nodular lymphocyte-predominant Hodgkin lymphoma)
* Indication for first-line systemic treatment with chemotherapy or chemoimmunotherapy
* Has signed the study-specific informed consent form
* Pre-treatment PET-CT scan performed
* Patient is affiliated with or a beneficiary of a health insurance plan

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient who has already started first-line chemotherapy or chemoimmunotherapy for lymphoma treatment (prephase corticosteroid therapy is allowed)
* Patient enrolled in a clinical trial evaluating an early-phase therapeutic agent (Phase I-II)
* Patient weighing less than 30 kg
* Adult under legal protection measures
* Patient unable to understand the study for any reason or unable to comply with the trial requirements (e.g., language barrier, psychological, or geographic issues).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the diagnostic performance of minimal residual disease (MRD) at the end of treatment in terms of sensitivity, specificity, positive predictive value, and negative predictive value for predicting 1-year progression-free survival (PFS). | 1 year
  Comparison with the diagnostic performance of PET-CT imaging at the end of first-line treatment for predicting 1-year PFS

SECONDARY OUTCOMES:
Response rates | 6 months
  Evaluation of responses based on PET-CT with Lugano 2014 Criteria
Overall survival | one year
  Time between inclusion and death

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Jacques Monod, Montivilliers
  - Centre Henri Becquerel, Rouen